CLINICAL TRIAL: NCT05723068
Title: Burden of Hepatitis D Virus (HDV) Infection in Italy: a Prospective/Observational Multicenter Study to Define Demographic, Clinical and Virological Features
Brief Title: Burden of Hepatitis D Virus (HDV) Infection in Italy
Acronym: HDV Describe
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IN-IT-980-6382
Record Dates: First submitted 2023-01-11; First posted 2023-02-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hepatitis D
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis D

SUMMARY:
The circulation of the Hepatitis D Virus (HDV) has considerably diminished in Italy, secondary to the control of the Hepatitis B Virus (HBV) with vaccination; this has led to the perception that HDV is vanishing and has reduced attention to the diagnosis of Hepatitis D. However, migratory fluxes from HDV endemic areas, fostered by labour-forces globalization, are increasingly reconstituting the reservoir of HDV in the country and hepatitis D has not yet vanished in native Italians but will remain an important medical issue for several years to come. As the epidemiologic and clinical features of HDV infection in migrant communities are largely unknown and the features of native Italians with long standing HDV infections have not been updated, this project intends to establish the contemporary epidemiological and medical context of HDV in immigrants in Italy and to determine the clinical characteristics and needs of the residual cohort of native HDV Italians, through the analysis of all HDV cases recruited in 12 months in a coordinated network of 35 Italian medical centers. The data will provide an appraisal of the burden of hepatitis D in the country and of its impact on the National Health System. They will present the paradigm of the current trend of HDV infection in high-income countries in the world.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positive subjects
* 18 years or older
* anti-HD-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in a Country-wide coordinated network of national medical centers. The network will include hepatology, infectious disease and internal medicine centers that historically care for patients with viral liver disease, located in the 12 major regions of Italy.
Sampling Method: Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics of HDV-infected patients | 1 year
  Demographic characteristics: age, sex, height, weight, nationality. HDV means hepatitis D virus
Epidemiologic characteristics of HDV-infected patients | 1 year
  Risk factors for infection. HDV means hepatitis D virus
Serum alanine aminotransferase concentration values in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Blood platelet count in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Serum albumin concentration values in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Serum total bilirubin concentration values in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Serum anti-liver-kidney microsomal antibodies titer in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Proportion of patients with detectable HDV RNA among seropositive anti-HDV patients | 1 year
  HDV means hepatitis D virus
Serum HDV RNA levels in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Proportion of HDV genotypes among patients with detectable HDV RNA | 1 year
  HDV means hepatitis D virus
Proportion of patients with detectable HBV DNA among seropositive anti-HDV | 1 year
  HBV means hepatitis B virus. HDV means hepatitis D virus
Serum HBV DNA levels in HDV-infected patients | 1 year
  HBV means hepatitis B virus. HDV means hepatitis D virus
Proportion of HBV genotypes among patients with detectable HBV DNA | 1 year
  HBV means hepatitis B virus
HBsAg concentration levels in HDV-infected patients | 1 year
  HBsAg means hepatitis B surface antigen. HDV means hepatitis D virus
HBcrAg concentration levels in HDV-infected patients | 1 year
  HBcrAg means hepatitis B core-related antigen. HDV means hepatitis D virus
Proportion of patients with liver cirrhosis among seropositive anti-HDV | 1 year
  HDV means hepatitis D virus
Liver stiffness values in HDV-infected patients | 1 year
  HDV means hepatitis D virus
Proportion of patients with hepatocellular carcinoma among seropositive anti-HDV | 1 year
  HDV means hepatitis D virus
Proportion of patients treated with antiviral therapy among seropositive anti-HDV | 1 year
  HDV means hepatitis D virus

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rizzetto, MD, Principal Investigator — University of Turin, Italy
Locations (36):
- Italy (36):
  - Università degli Studi di Bari Aldo Moro, Bari
  - Gastroenterology Hepatology and Transplantation, ASST Bergamo, Bergamo
  - Malattie Infettive, ASST Bergamo, Bergamo
  - Dipartimento di Scienze Mediche e Chirurgiche, Università degli Studi di Bologna, Bologna
  - Dipartimento di Scienze Cliniche e Sperimentali, Università degli Studi di Brescia, Brescia
  - UOC Malattie Infettive e Tropicali, A.O. S Anna e S Sebastiano, Caserta
  - UOS Epatologia "G. Rodolico-San Marco", Catania
  - UOC Medicina Interna Ospedaliera, Policlinico "Mater Domini", Catanzaro
  - Dipartimento di Medicina Clinica e Sperimentale, Università degli Studi di Foggia, Foggia
  - S.C. Malattie Infettive, E.O. Ospedali Galliera, Genova
  - UOC Malattie Infettive, Ospedale Paolo Borsellino di Marsala, Marsala
  - A.O.U. Policlinico G. Martino di Messina, Università di Messina, Messina
  - Dipartimento di Malattie Infettive e Centro Epatopatie, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Dipartimento di Malattie Infettive, ASST Fatebenefratelli - Ospedale Luigi Sacco, Milan
  - UOC Gastroenterologia e Epatologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Università degli Studi di Milano, Milan
  - UOC di Medicina Interna Metabolica, AOU di Modena e Università di Modena e Reggio, Modena
  - Dipartimento di Malattie Infettive, Ospedale D. Cotugno, Napoli
  - Dipartimento di Medicina di Precisione, Università della Campania "Luigi Vanvitelli", Napoli
  - Dipartimento di Medicina e Chirurgia, Università degli Studi di Napoli Federico II, Napoli
  - Dipartimento di Medicina Interna, Università della Campania "Luigi Vanvitelli", Napoli
  - Dipartimento di Medicina Traslazionale, Università del Piemonte Orientale, Novara
  - UOC Malattie Infettive e Tropicali, Azienda Ospedale-Università di Padova, Padua
  - Dipartimento di Promozione della Salute, Materno-Infantile di Medicina Interna e Specialistica di Eccellenza "G. D'Alessandro", Università degli Studi di Palermo, Palermo
  - UOC di Malattie Infettive, Università di Parma, Parma
  - Dipartimento di Medicina Clinica e Sperimentale, Università di Pisa, Pisa
  - UOC Malattie Infettive, Grande Ospedale Metropolitano "Bianchi - Melacrino - Morelli", Reggio Calabria
  - Malattie Infettive Roma 2, Roma
  - Ospedale S. Andrea, Roma
  - Policlinico Gemelli, Roma
  - UOC Malattie Infettive Epatologia, IRCCS Lazzaro Spallanzani, Roma
  - Unità di Gastroenterologia ed Endoscopia Digestiva, IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - UOC Malattie Infettive, Syracuse
  - Clinica Universitaria Malattie Infettive, Ospedale Amedeo di Savoia, Torino
  - Unit of Gastroenterology, University of Turin, Torino
  - Unità di Epatologia e Trapianti di Fegato, Università degli Studi di Udine, Udine
  - UO Malattie Infettive, Azienda Ospedaliera Universitaria Integrata Verona, Verona

IPD SHARING:
Plan to Share IPD: No